CLINICAL TRIAL: NCT07281378
Title: Reducing Co-occurring Substance Use and HIV Risk Among Stimulant-using Men at High Risk for HIV in the United States of America.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB202501242; 5R00DA053158-05 (NIH)
Record Dates: First submitted 2025-12-11; First posted 2025-12-15 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-10

CONDITIONS: Drug Use Disorders; PrEP Uptake; PrEP Adherence; HIV Risk Behavior
Keywords: PrEP; PrEP uptake; HIV; substance use; stimulant use; men at high risk for HIV
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention-Control condition (Other): Participants randomized to the control condition will have six 1-on-1 sessions with a facilitator engaging in writing exercises. The sessions will be comparable in length to the intervention sessions but will not include any skills practice. Each session will include a neutral writing exercises.
  Interventions: Behavioral: Contingency Management
- Experimental condition (Experimental): Participants randomized to the experimental condition (tailored behavioral intervention) will have a 1-on-1 session with a facilitator. The intervention consists of six individually delivered sessions (1-2 sessions per week, approximately 1.5 hours each). The intervention will be interactive and include rapport- and trust-building activities; didactic teaching; multimedia (e.g., videos) messages to facilitate modeling and discussion; role-playing and skills building, practice, and feedback. The intervention will be led by a CITI certified facilitator, who is also a member of the study team. The sessions are: (1) Positive affect skills; (2) Positive Conscious Networks broaden and building supportive personal networks; (3) Mindfulness; (4) Personal Strengths and Obtainable Goals; (5) Positive Reassessment; and (6) Compassion/solidarity to one-self as to others. Sessions/modules will be guided by Segmented Assimilation and Stress and Coping Theory.
  Interventions: Behavioral: Tailored Positive Affect Intervention; Behavioral: Contingency Management

INTERVENTIONS:
Behavioral: Tailored Positive Affect Intervention — The intervention consists of six individually delivered sessions (1-2 sessions per week, approximately 1.5 hours each). The intervention will be interactive and include rapport- and trust-building activities; didactic teaching; multimedia (e.g., videos) messages to facilitate modeling and discussion; role-playing and skills building, practice, and feedback. T
  The sessions are: (1) Positive affect skills; (2) Positive Conscious Networks broaden and building supportive personal networks;(3) Mindfulness; (4) Personal Strengths and Obtainable Goals; (5) Positive Reassessment; and (6) Compassion/solidarity to one-self as to others. Sessions/modules will be guided by Segmented Assimilation and Stress and Coping Theory.
  Arms: Experimental condition
Behavioral: Contingency Management — Incentives will be provided as positive reinforcement of two key behaviors that are crucial to increase PrEP uptake. First, participants will receive incentives for documented evidence that they have completed a medical visit for PrEP clinical evaluation (including HIV testing). Second, participants completing PrEP clinical evaluation will receive incentives when they document evidence of an active prescription of PrEP.

SUMMARY:
This intervention will focus on stimulant-using men at high risk for HIV who are in need of tailored behavioral interventions to mitigate co-occurring stimulant use and HIV risk in the era of pre-exposure prophylaxis (PrEP). The study is a pilot randomized controlled trial to evaluate the adaptation, feasibility, acceptability, and preliminary efficacy of a behavioral intervention.

ELIGIBILITY:
Inclusion Criteria:

1. be 18 years of age or older;
2. be sexually active cisgender men at high risk for HIV (foreign and US-born, residing in the US)-reporting any condomless anal sex (CAS) in the past three months with a man;
3. report use of stimulant (i.e., methamphetamine, powder cocaine, or crack-cocaine) at least one day in the past three or six month;
4. have HIV-negative serostatus;
5. be bilingual (Spanish and English), or Spanish or English monolingual;
6. meet CDC criteria for PrEP eligibility.

Exclusion Criteria:

1. display diminished capacity to consent (e.g., cognitive impairment); or
2. severe psychiatric symptoms (e.g., psychosis) that require more intensive treatment;
3. if they are HIV positive or living with HIV;
4. if they are already taking PrEP; and
5. if the participant can't consent to participate in English or Spanish.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender men
Enrollment: 84 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of PrEP uptake | From enrollment to 6 months
  Changes in number of participants obtaining prescription to begin PrEP. Measured through documented evidence of an active prescription for PrEP.

SECONDARY OUTCOMES:
Stimulant use (self-report) | Enrollment to 6 months
  Changes in the severity of participant stimulant use as measured by the Alcohol, Smoking, and Substance Involvement Screen Test (ASSIST) composite scores for cocaine and amphetamine-type stimulants.
Condomless Anal Sex (CAS) | From enrollment to 6 months
  Changes in the number of CAS partners who are not taking PrEP or virally suppressed.
Social Network Composition | From enrollment to 6 months
  Changes in the number of social network alters who use stimulants and increases in the number of social network alters who are taking PrEP.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Colon-Burgos, DrPH, Principal Investigator — University of Florida

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets from the study will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: 12 months after completion of the study
Access Criteria: Data will be accessible via UF data repository

REFERENCES:
- [Background] Cohen J. Statistical Power Analysis for the Behavioral Sciences. 2nd ed. Hillsdale, New Jersey: Lawrence Earlbaum Associates; 1988.
- [Background] Kraemer HC, Wilson GT, Fairburn CG, Agras WS. Mediators and moderators of treatment effects in randomized clinical trials. Arch Gen Psychiatry. 2002 Oct;59(10):877-83. doi: 10.1001/archpsyc.59.10.877. PMID 12365874
- [Background] Molenberghs G, Verbeke G. Models for Discrete Longituidnal Data. New York: Springer- Verlag; 2005.
- [Background] Reback CJ, Peck JA, Dierst-Davies R, Nuno M, Kamien JB, Amass L. Contingency management among homeless, out-of-treatment men who have sex with men. J Subst Abuse Treat. 2010 Oct;39(3):255-63. doi: 10.1016/j.jsat.2010.06.007. Epub 2010 Jul 29. PMID 20667681
- [Background] Shoptaw S, Reback CJ, Peck JA, Yang X, Rotheram-Fuller E, Larkins S, Veniegas RC, Freese TE, Hucks-Ortiz C. Behavioral treatment approaches for methamphetamine dependence and HIV-related sexual risk behaviors among urban gay and bisexual men. Drug Alcohol Depend. 2005 May 9;78(2):125-34. doi: 10.1016/j.drugalcdep.2004.10.004. Epub 2004 Nov 28. PMID 15845315
- [Background] Shoptaw S, Klausner JD, Reback CJ, Tierney S, Stansell J, Hare CB, Gibson S, Siever M, King WD, Kao U, Dang J. A public health response to the methamphetamine epidemic: the implementation of contingency management to treat methamphetamine dependence. BMC Public Health. 2006 Aug 18;6:214. doi: 10.1186/1471-2458-6-214. PMID 16919170
- [Background] Saldaña J. The Coding Manual for Qualitative Researchers. 3rd ed. Los Angeles, CA: SAGE; 2016.
- [Background] Creswell JW. Qualitative Inquiry and Research Design: Choosing among Five Approaches. 3ed ed. Thousand Oaks,California: SAGE Publications; 2013.
- [Background] Centers for Disease Control and Prevention. Preexposure Prophylaxis for the Prevention of HIV Infection in the United States - 2017 Clinical Practice Guideline.; 2018. https://www.cdc.gov/std/tg2015/tg-2015-.
- [Background] Mccarty C, Lubbers MJ, Vacca R, Molina JL. Conducting Personal Network Research: A Practical Guide. New York, N.Y.: The Guilford Press; 2019. www.guilford.com.
- [Background] 27855594
- [Background] Padilla M, Colon-Burgos JF, Varas-Diaz N, Matiz-Reyes A, Parker CM. Tourism Labor, Embodied Suffering, and the Deportation Regime in the Dominican Republic. Med Anthropol Q. 2018 Dec;32(4):498-519. doi: 10.1111/maq.12447. Epub 2018 May 8. PMID 29665064
- [Background] Colon Burgos JF, Padilla M, Nunez A, Varas-Diaz N, Matiz-Reyes A. An ethnographic study of 'touristic escapism' and health vulnerability among Dominican male tourism workers. Glob Public Health. 2019 Nov;14(11):1578-1588. doi: 10.1080/17441692.2019.1651370. Epub 2019 Aug 9. PMID 31397201
- [Background] Carrico AW, Zepf R, Meanley S, Batchelder A, Stall R. Critical Review: When the Party is Over: A Systematic Review of Behavioral Interventions for Substance-Using Men Who Have Sex with Men. J Acquir Immune Defic Syndr. 2016 Nov 1;73(3):299-306. doi: 10.1097/QAI.0000000000001102. PMID 27258233
- [Background] Folkman S. The case for positive emotions in the stress process. Anxiety Stress Coping. 2008 Jan;21(1):3-14. doi: 10.1080/10615800701740457. PMID 18027121
- [Background] Carrico AW, Neilands TB, Dilworth SE, Evans JL, Gomicronmez W, Jain JP, Gandhi M, Shoptaw S, Horvath KJ, Coffin L, Discepola MV, Andrews R, Woods WJ, Feaster DJ, Moskowitz JT. Randomized controlled trial of a positive affect intervention to reduce HIV viral load among sexual minority men who use methamphetamine. J Int AIDS Soc. 2019 Dec;22(12):e25436. doi: 10.1002/jia2.25436. PMID 31860172
- [Background] Bernal G, Saez-Santiago E. Culturally Centered Psychosocial Interventions. Focus (Am Psychiatr Publ). 2024 Oct;22(4):508-514. doi: 10.1176/appi.focus.24022022. Epub 2024 Oct 15. PMID 39563877
- [Background] Akresh IR, Do DP, Frank R. Segmented assimilation, neighborhood disadvantage, and Hispanic immigrant health. Soc Sci Med. 2016 Jan;149:114-21. doi: 10.1016/j.socscimed.2015.12.013. Epub 2015 Dec 13. PMID 26708247
- [Background] Garcia M, Harris AL. PrEP awareness and decision-making for Latino MSM in San Antonio, Texas. PLoS One. 2017 Sep 27;12(9):e0184014. doi: 10.1371/journal.pone.0184014. eCollection 2017. PMID 28953905
- [Background] Brooks RA, Nieto O, Landrian A, Fehrenbacher A, Cabral A. Experiences of Pre-Exposure Prophylaxis (PrEP)-Related Stigma among Black MSM PrEP Users in Los Angeles. J Urban Health. 2020 Oct;97(5):679-691. doi: 10.1007/s11524-019-00371-3. PMID 31214977
- [Background] Castro FG, Marsiglia FF, Kulis S, Kellison JG. Lifetime segmented assimilation trajectories and health outcomes in Latino and other community residents. Am J Public Health. 2010 Apr;100(4):669-76. doi: 10.2105/AJPH.2009.167999. Epub 2010 Feb 18. PMID 20167890
- [Background] Sauceda JA, Brooks RA, Xavier J, Maiorana A, Georgetti Gomez L, Zamudio-Haas S, Rodriguez-Diaz CE, Cajina A, Myers J. From Theory to Application: A Description of Transnationalism in Culturally-Appropriate HIV Interventions of Outreach, Access, and Retention Among Latino/a Populations. J Immigr Minor Health. 2019 Apr;21(2):332-345. doi: 10.1007/s10903-018-0753-2. PMID 29767401
- [Background] Centers for Disease Control and Prevention. Estimated HIV Incidence and Prevalence in the United States, 2010-2016. Vol 24. Atlanta, Georgia; 2019. http://www.cdc.gov/hiv/library/reports/hivsurveillance. html.http://www.cdc.gov/hiv/library/reports/hivsurveillance. htmlhttp://wwwn.cdc.gov/dcs/ContactUs/Form.
- [Background] Brooks RA, Nieto O, Landrian A, Donohoe TJ. Persistent stigmatizing and negative perceptions of pre-exposure prophylaxis (PrEP) users: implications for PrEP adoption among Latino men who have sex with men. AIDS Care. 2019 Apr;31(4):427-435. doi: 10.1080/09540121.2018.1499864. Epub 2018 Jul 18. PMID 30021456
- [Background] Rhodes SD, McCoy TP, Vissman AT, DiClemente RJ, Duck S, Hergenrather KC, Foley KL, Alonzo J, Bloom FR, Eng E. A randomized controlled trial of a culturally congruent intervention to increase condom use and HIV testing among heterosexually active immigrant Latino men. AIDS Behav. 2011 Nov;15(8):1764-75. doi: 10.1007/s10461-011-9903-4. PMID 21301948
- [Background] Perez A, Santamaria EK, Operario D. A Systematic Review of Behavioral Interventions to Reduce Condomless Sex and Increase HIV Testing for Latino MSM. J Immigr Minor Health. 2018 Oct;20(5):1261-1276. doi: 10.1007/s10903-017-0682-5. PMID 29247266
- [Background] Rhodes SD, McCoy TP, Hergenrather KC, Vissman AT, Wolfson M, Alonzo J, Bloom FR, Alegria-Ortega J, Eng E. Prevalence estimates of health risk behaviors of immigrant latino men who have sex with men. J Rural Health. 2012 Jan;28(1):73-83. doi: 10.1111/j.1748-0361.2011.00373.x. Epub 2011 Mar 31. PMID 22236317
- [Background] Fernandez MI, Jacobs RJ, Warren JC, Sanchez J, Bowen GS. Drug use and Hispanic men who have sex with men in South Florida: implications for intervention development. AIDS Educ Prev. 2009 Oct;21(5 Suppl):45-60. doi: 10.1521/aeap.2009.21.5_supp.45. PMID 19824834
- [Background] Fernandez MI, Bowen GS, Varga LM, Collazo JB, Hernandez N, Perrino T, Rehbein A. High rates of club drug use and risky sexual practices among Hispanic men who have sex with men in Miami, Florida. Subst Use Misuse. 2005;40(9-10):1347-62. doi: 10.1081/JA-200066904. PMID 16048821
- [Background] Egan JE, Frye V, Kurtz SP, Latkin C, Chen M, Tobin K, Yang C, Koblin BA. Migration, neighborhoods, and networks: approaches to understanding how urban environmental conditions affect syndemic adverse health outcomes among gay, bisexual and other men who have sex with men. AIDS Behav. 2011 Apr;15 Suppl 1(Suppl 1):S35-50. doi: 10.1007/s10461-011-9902-5. PMID 21369730
- [Background] Finlayson TJ, Le B, Smith A, Bowles K, Cribbin M, Miles I, Oster AM, Martin T, Edwards A, Dinenno E; Centers for Disease Control and Prevention (CDC). HIV risk, prevention, and testing behaviors among men who have sex with men--National HIV Behavioral Surveillance System, 21 U.S. cities, United States, 2008. MMWR Surveill Summ. 2011 Oct 28;60(14):1-34. PMID 22031280
- [Background] NDEWS. Methamphetamine Highlights.; 2018. https://ndews.umd.edu/sentinelsites/ sentinel-sites-reports-and-community-contacts.
- [Background] Oldenburg CE, Jain S, Mayer KH, Mimiaga MJ. Post-exposure prophylaxis use and recurrent exposure to HIV among men who have sex with men who use crystal methamphetamine. Drug Alcohol Depend. 2015 Jan 1;146:75-80. doi: 10.1016/j.drugalcdep.2014.11.010. Epub 2014 Nov 26. PMID 25482500
- [Background] Plankey MW, Ostrow DG, Stall R, Cox C, Li X, Peck JA, Jacobson LP. The relationship between methamphetamine and popper use and risk of HIV seroconversion in the multicenter AIDS cohort study. J Acquir Immune Defic Syndr. 2007 May 1;45(1):85-92. doi: 10.1097/QAI.0b013e3180417c99. PMID 17325605
- [Background] Koblin BA, Husnik MJ, Colfax G, Huang Y, Madison M, Mayer K, Barresi PJ, Coates TJ, Chesney MA, Buchbinder S. Risk factors for HIV infection among men who have sex with men. AIDS. 2006 Mar 21;20(5):731-9. doi: 10.1097/01.aids.0000216374.61442.55. PMID 16514304
- [Background] Ostrow DG, Plankey MW, Cox C, Li X, Shoptaw S, Jacobson LP, Stall RC. Specific sex drug combinations contribute to the majority of recent HIV seroconversions among MSM in the MACS. J Acquir Immune Defic Syndr. 2009 Jul 1;51(3):349-55. doi: 10.1097/QAI.0b013e3181a24b20. PMID 19387357
- [Background] Portes A, Zhou M. The New Second Generation : Segmented Assimilation and its Variants. Ann Am Acad Pol Soc Sci. 1993;530:74-96.
- [Background] Bernal G, Bonilla J, Bellido C. Ecological validity and cultural sensitivity for outcome research: issues for the cultural adaptation and development of psychosocial treatments with Hispanics. J Abnorm Child Psychol. 1995 Feb;23(1):67-82. doi: 10.1007/BF01447045. PMID 7759675
- [Background] Folkman S, Moskowitz JT. Positive affect and the other side of coping. Am Psychol. 2000 Jun;55(6):647-54. doi: 10.1037//0003-066x.55.6.647. PMID 10892207
- [Background] Carrico AW, Gomicronmez W, Jain J, Shoptaw S, Discepola MV, Olem D, Lagana-Jackson J, Andrews R, Neilands TB, Dilworth SE, Evans JL, Woods WJ, Moskowitz JT. Randomized controlled trial of a positive affect intervention for methamphetamine users. Drug Alcohol Depend. 2018 Nov 1;192:8-15. doi: 10.1016/j.drugalcdep.2018.07.029. Epub 2018 Sep 5. PMID 30195243
- [Background] Kelly JA, Amirkhanian YA, Seal DW, Galletly CM, Difranceisco W, Glasman LR, Stevenson LY, Rosado N. Levels and Predictors of Sexual HIV Risk in Social Networks of Men who Have Sex with Men in the Midwest. AIDS Educ Prev. 2010 Dec;22(6):483-95. doi: 10.1521/aeap.2010.22.6.483. PMID 21204625
- [Background] Sanchez M, Dillon FR, Concha M, De La Rosa M. The Impact of Religious Coping on the Acculturative Stress and Alcohol Use of Recent Latino Immigrants. J Relig Health. 2015 Dec;54(6):1986-2004. doi: 10.1007/s10943-014-9883-6. PMID 24859922
- [Background] Colon-Burgos J, Padilla MB, Buttram M, Varas N. Examining the syndemic of drug use and HIV among Latino MSM that work in the tourism sector of South Beach. In: American Public Health Association; 2019.
- [Background] Hojilla JC, Vlahov D, Crouch PC, Dawson-Rose C, Freeborn K, Carrico A. HIV Pre-exposure Prophylaxis (PrEP) Uptake and Retention Among Men Who Have Sex with Men in a Community-Based Sexual Health Clinic. AIDS Behav. 2018 Apr;22(4):1096-1099. doi: 10.1007/s10461-017-2009-x. PMID 29243109
- [Background] Lewis NM, Wilson K. HIV risk behaviours among immigrant and ethnic minority gay and bisexual men in North America and Europe: A systematic review. Soc Sci Med. 2017 Apr;179:115-128. doi: 10.1016/j.socscimed.2017.02.033. Epub 2017 Feb 24. PMID 28260636
- [Background] Hojilla JC, Vlahov D, Glidden DV, Amico KR, Mehrotra M, Hance R, Grant RM, Carrico AW. Skating on thin ice: stimulant use and sub-optimal adherence to HIV pre-exposure prophylaxis. J Int AIDS Soc. 2018 Mar;21(3):e25103. doi: 10.1002/jia2.25103. PMID 29577616
- [Background] Hojilla JC, Satre DD, Glidden DV, McMahan VM, Gandhi M, Defechereux P, Guanira JV, Mehrotra M, Grant RM, Carrico AW. Brief Report: Cocaine Use and Pre-exposure Prophylaxis: Adherence, Care Engagement, and Kidney Function. J Acquir Immune Defic Syndr. 2019 May 1;81(1):78-82. doi: 10.1097/QAI.0000000000001972. PMID 30730359
- [Background] CDC. Diagnoses of HIV Infection in the United States and Dependent Areas, 2018 (Preliminary) HIV Surveillance Supplemental Report 2 Vol. 30. Atlanta, Georgia; 2019. http://www.cdc.gov/hiv/library/reports/hivsurveillance. html.http://www.cdc.gov/hiv/library/reports/hivsurveillance. htmlhttp://wwwn.cdc.gov/dcs/ContactUs/Form.
- [Background] Rhodes SD, Alonzo J, Mann L, Freeman A, Sun CJ, Garcia M, Painter TM. Enhancement of a Locally Developed HIV Prevention Intervention for Hispanic/Latino MSM: A Partnership of Community-Based Organizations, a University, and the Centers for Disease Control and Prevention. AIDS Educ Prev. 2015 Aug;27(4):312-32. doi: 10.1521/aeap.2015.27.4.312. PMID 26241382
- [Background] U.S. Department of Health & Human Services. What is 'Ending the HIV Epidemic: A Plan for America'? | HIV.gov. https://www.hiv.gov/federal-response/ending-the-hivepidemic/ overview.